CLINICAL TRIAL: NCT00128141
Title: Effect of Maternal Tactile and Kinesthetic Stimulation on Length of Hospital Stay of Very Low Birth Weight Infants
Brief Title: Effect of Tactile and Kinesthetic Stimulation on Very Low Birth Weight Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Bioethics Commission of Brazil (Other)
Responsible Party: Renato S. Procianoy, Hospital de Clinicas de Porto Alegrte
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HCPA03287
Record Dates: First submitted 2005-08-08; First posted 2005-08-09 (Estimated); Last update posted 2008-02-05 (Estimated); Status verified 2008-02

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth | interventions — Massage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention)
- 2 (Experimental): tactile stimulus
  Interventions: Behavioral: Tactile stimulus

INTERVENTIONS:
Behavioral: Tactile stimulus — four times a day
  Other Names: massage therapy
  Arms: 2

SUMMARY:
Two groups of preterm infants with birth weight equal to or less than 1500 grams will be studied. One group will receive the standard care and the other will receive standard care plus maternal special tactile stimulation. Gain of weight, length and head circumference, date of the beginning of enteral feedings, length of time to recover birth weight and age of hospital discharge will be recorded and compared between both groups.

DETAILED DESCRIPTION:
Preterm infants birth weight equal or less than 1500 grams and gestational age equal or less than 32 weeks will be randomized in two groups: standard care that will receive the usual treatment applied to all infants admitted to our unit and a second groups that will receive standard care plus maternal tactile and kinesthetic stimuli that will be taught to the mothers. Randomization will be performed among those that accept to participate in the study. Growth (birth, length and head circumference), age of life to start receiving enteral feedings, length of hospital stay, time to recover birth weight will be recorded and compared between both groups.

ELIGIBILITY:
Inclusion Criteria:

* Preterm newborns with birth weight equal to or less than 1500 grams and gestational age equal to or less than 32 weeks.
* Mother willing to participate in study.

Exclusion Criteria:

* Major congenital malformations
* Congenital infectious diseases
* Mother not willing to participate in study

Ages: 1 Hour to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2003-08; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
length of hospital stay

SECONDARY OUTCOMES:
effect on beginning of enteral feedings
growth during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Renato S Procianoy, MD, Principal Investigator — Universidade Federal do Rio Grande do Sul-Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil